CLINICAL TRIAL: NCT01687985
Title: A Safety and Efficacy Evaluation of BLI801 Laxative in Constipated Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BLI801-202
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BLI801 laxative - low dose (Experimental): BLI801 laxative - oral solution
  Interventions: Drug: BLI801 laxative - low dose
- BLI801 laxative - high dose (Experimental): BLI801 laxative - oral solution
  Interventions: Drug: BLI801 laxative - high dose

INTERVENTIONS:
Drug: BLI801 laxative - low dose — BLI801 laxative - oral solution
  Arms: BLI801 laxative - low dose
Drug: BLI801 laxative - high dose — BLI801 laxative - oral solution
  Other Names: BLI801
  Arms: BLI801 laxative - high dose

SUMMARY:
A pilot study to evaluate the safety and efficacy of multiple BLI801 doses in constipated adults.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects at least 18 years of age

Constipated, defined by ROME definition:

Otherwise in good health, as determined by physical exam and medical history

Exclusion Criteria:

Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon

Subjects taking laxatives or prokinetic agents that refuse to discontinue these treatments

Subjects who are allergic to any BLI801 component

Subjects currently taking narcotic analgesics or other medications known to cause constipation

Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures

Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days

Subjects with an active history of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Treatment Success | 4 weeks
  percent of patients experiencing a response in 3 out of 4 weeks of treatment

SECONDARY OUTCOMES:
serum chemistry | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, Anaheim, California
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Clinsearch, Chattanooga, Tennessee
  - Memphis Gastroenterology, Germantown, Tennessee